CLINICAL TRIAL: NCT03974087
Title: The Effect of Transcranial Direct Current Stimulation on Visual Attention in Mild Cognitive Impairment - a Combined MRI and Non-invasive Brain Stimulation Study
Brief Title: The Effect of Transcranial Direct Current Stimulation on Visual Attention in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NV18-04-00256
Record Dates: First submitted 2019-05-10; First posted 2019-06-04 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2021-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Transcranial direct current stimulation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCI patients with real transcranial direct current stimulation (Active Comparator): Patients will receive 2mA stimulation in 10 consecutive sessions.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- MCI patients with sham transcranial direct current stimulation (Sham Comparator): Patients will receive sham stimulation in 10 consecutive sessions.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — 2mA stimulation for 20 minutes

SUMMARY:
Progressively causes the breakdown of cognitive functions and impairs quality of life for patients and their caregivers. In addition to memory impairment, visual attention is also compromised, even at the stage of mild cognitive impairment due to AD (MCI-AD). No treatment has been found for MCI-AD; therefore, attention has been drawn to non-invasive brain stimulation techniques, such as transcranial direct current stimulation (tDCS), in order to enhance cognitive functions by modifying brain plasticity. In the current research, investigator aim to examine the long-term effects of the optimal multiple-session tDCS protocol in MCI-AD on visual attention including the transfer to an ecologically valid virtual environment and identify the neural underpinnings of tDCS-induced behavioral aftereffects using a combined tDCS/ MRI network-based approach.

DETAILED DESCRIPTION:
Investigator will investigate the long-term effects of 10 active tDCS consecutive sessions using an optimized stimulation protocol as compared to a placebo stimulation on visual attention in the MCI-AD. A two-parallel-group, randomized, placebo-controlled design will be used. In addition, the cognitive transfer of tDCS will be evaluated. Repeated tDCS sessions will be performed in 10 consecutive sessions (2 weeks: Monday to Friday) over one preselected ROI together with ongoing visual attention training. During the stimulation, investigator will use the visual matching task. Before the repeated stimulation sessions, participants will undergo the neurocognitive examination. Behavioral examinations of the trained and untrained tasks (i.e. the transfer tasks) will be performed to assess the baseline performance. MRI protocol consisting of T1, T2, FLAIR, and fMRI during the task performance (visual matching task), resting state fMRI, and DTI sequences will be acquired before and after the whole 10-day stimulation protocol in order to search for active vs. placebo tDCS-induced changes in brain activation and resting state functional and structural connectivity and to identify neural correlates of behavioral changes. Behavioral assessment of the trained task and the transfer task will be repeated immediately after and again at a one-month follow-up visit after the end of the last stimulation session

ELIGIBILITY:
Inclusion Criteria:

* amnestic single or multi-domain mild cognitive impairment patients in accordance with diagnostic criteria (Albert et al., 2011)

Exclusion Criteria:

* psychiatric disorders, including major depression, major vascular lesions, and other brain pathologies detected by MRI that might present with cognitive decline
* a cardio pacemaker or any MRI-incompatible metal in the body
* epilepsy
* any diagnosed psychiatric disorder
* alcohol/drug abuse
* lack of cooperation
* presence of dementia.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Visual-attention task accuracy | Change from baseline immediately after completion of stimulation protocol and one month after completion of stimulation protocol
  Task will be presented on a computer and subject will respond by YES-NO buttons. Only if there are no differences in task accuracy, we will measure task reaction times (e.g. due to the roof effect).

SECONDARY OUTCOMES:
Psychological assessment - z-score computed from multiple psychological domains | Change from baseline immediately after one month from completion of stimulation protocol
  Z-scores based on neuropsychological assessment (lasting up to 40 min) evaluating (global cognitive functions, memory, attention, psychomotor functions, executive functions, visuospatial functions, language, depressive symptoms, and activities of daily living) Only if there are no changes in z-score, we will asses change on a level of individual tests.
Magnetic resonance imaging | Change from baseline immediately after completion of stimulation protocol and one month after completion of stimulation protocol
  Investigator will record high resolution structural T1-weighted (MPRAGE) images, functional T2* weighted multiband EPI sequences, and DTI measurement. The total time spent in the scanner will be approximately 60 min

OTHER OUTCOMES:
Memory task in virtual reality performance - the accuracy | Change from baseline immediately after completion of stimulation protocol and one month after completion of stimulation protocol
Memory task in virtual reality performance - The time to accomplish different difficulty levels | Change from baseline immediately after completion of stimulation protocol and one month after completion of stimulation protocol
Memory task in virtual reality performance - The trajectories needed for completion of different difficulty levels | Change from baseline immediately after completion of stimulation protocol and one month after completion of stimulation protocol
Visual working memory task accuracy | Change from baseline immediately after completion of stimulation protocol and one month after completion of stimulation protocol
  Task will be presented on a computer and subject will respond by YES-NO buttons. Only if there are no differences in task accuracy, we will measure task reaction times (e.g. due to the roof effect).

CONTACTS AND LOCATIONS:
Overall Officials: Lubomira Anderková, PhD, Principal Investigator — Ceitec, Masaryk University
Locations (1):
- Ceitec, Masaryk University, Brno, Czechia